CLINICAL TRIAL: NCT03321942
Title: The Biological Characteristics of Adipose Tissue-derived Mesenchymal Stem Cells and Its Role in the Treatment of Chronic Renal Failure
Brief Title: Treatment of Chronic Renal Failure With Adipose Tissue-derived Mesenchymal Stem Cells
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Affiliated Hospital of Xuzhou Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: XYFY2016-KL031-01
Record Dates: First submitted 2017-10-19; First posted 2017-10-26 (Actual); Last update posted 2017-10-26 (Actual); Status verified 2017-10

CONDITIONS: Mesenchymal Stem Cells; Chronic Kidney Diseases; Renal Interstitial Fibrosis
Keywords: Adipose Tissue-derived Mesenchymal Stem Cells; Chronic Kidney Diseases
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment group (Active Comparator): Adipose tissue-derived mesenchymal stem cells were used to treat patients with chronic renal failure.
  Interventions: Drug: Treatment group
- Control group (Placebo Comparator): Treatment of chronic renal failure patients with conventional methods.
  Interventions: Drug: Control group

INTERVENTIONS:
Drug: Treatment group — Adipose tissue-derived mesenchymal stem cells were used to treat patients with chronic renal failure on the basis of conventional treatment.
  Other Names: Stem cells treatment group
  Arms: Treatment group
Drug: Control group — Conventional treatment were used to treat patients with chronic renal failure.
  Other Names: Conventional treatment group
  Arms: Control group

SUMMARY:
To investigate the biological characteristics of adipose tissue-derived mesenchymal stem cells(AMSCs) and its treatment effects on chronic renal failure.

DETAILED DESCRIPTION:
This study aims to investigate the biological characteristics of adipose tissue-derived mesenchymal stem cells(AMSCs) and its effect on oxidative stress, inflammation and mitochondrial damage.We intend to use blood oxygen level-dependent magnetic resonance imaging(BOLD-MRI), emission computed tomography(ECT) and enhanced magnetic resonance imaging to monitor renal oxygenation, tissue perfusion and renal function.Ultimately, we evaluate the treatment effects of AMSCs on chronic renal failure through these observations mentioned above.We hope to delay the progression of renal function in patients with chronic renal failure, and save huge social cost for dialysis by these research.

ELIGIBILITY:
Inclusion Criteria:

* Enroll the chronic renal failure patients without dialysis in the department of nephrology of Affiliated Hospital of Xuzhou Medical University from January 2017 to December 2018.
* The patients enrolled were not treated with drugs that affect the renal blood flow and oxygen consumption, such as ACEI, ARB, calcium channel blockers, diuretics, vasodilators and other related factors within 2 weeks.

Exclusion Criteria:

* Exclude those patients with diabetes, cardiovascular disease, severe infection, shock, dehydration, abnormal liver function, received glucocorticoid therapy, surgery and emergency dialysis.
* Eliminate those patients with respiratory disease(such as chronic obstructive pulmonary disease, bronchiectasis, asthma), cardiovascular diseases(such as acute and chronic cardiac insufficiency), blood system diseases (such as aplastic anemia, nutritional anemia and polycythemia vera).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2017-01-01 (Actual); Primary Completion 2018-12-31 (Estimated); Study Completion 2018-12-31 (Estimated)

PRIMARY OUTCOMES:
serum creatinine | after 3 months of adipose tissue-derived mesenchymal stem cells treatment
  intravenous blood sampling

SECONDARY OUTCOMES:
glomerular filtration rate | after 3 months of adipose tissue-derived mesenchymal stem cells treatment
  emission computed tomography
apparent relaxation rate | after 3 months of adipose tissue-derived mesenchymal stem cells treatment
  blood oxygen level dependent magnetic resonance imaging

CONTACTS AND LOCATIONS:
Overall Officials: Dong Sun, MD, Study Director — The Affiliated Hospital of Xuzhou Medical University
Locations (1):
- The Affiliated Hospital of Xuzhou Medical University, Xuzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tayebati SK, Tomassoni D, Di Cesare Mannelli L, Amenta F. Effect of treatment with the antioxidant alpha-lipoic (thioctic) acid on heart and kidney microvasculature in spontaneously hypertensive rats. Clin Exp Hypertens. 2016;38(1):30-8. doi: 10.3109/10641963.2015.1047950. Epub 2015 Jul 24. PMID 26207883
- [Background] Prasad GV. Metabolic syndrome and chronic kidney disease: Current status and future directions. World J Nephrol. 2014 Nov 6;3(4):210-9. doi: 10.5527/wjn.v3.i4.210. PMID 25374814
- [Background] Maugeri N, Rovere-Querini P, Baldini M, Baldissera E, Sabbadini MG, Bianchi ME, Manfredi AA. Oxidative stress elicits platelet/leukocyte inflammatory interactions via HMGB1: a candidate for microvessel injury in sytemic sclerosis. Antioxid Redox Signal. 2014 Mar 1;20(7):1060-74. doi: 10.1089/ars.2013.5298. Epub 2014 Jan 17. PMID 24070090
- [Background] Sun D, Eirin A, Zhu XY, Zhang X, Crane JA, Woollard JR, Lerman A, Lerman LO. Experimental coronary artery stenosis accelerates kidney damage in renovascular hypertensive swine. Kidney Int. 2015 Apr;87(4):719-27. doi: 10.1038/ki.2014.343. Epub 2014 Oct 22. PMID 25337776
- [Background] Eirin A, Ebrahimi B, Zhang X, Zhu XY, Woollard JR, He Q, Textor SC, Lerman A, Lerman LO. Mitochondrial protection restores renal function in swine atherosclerotic renovascular disease. Cardiovasc Res. 2014 Sep 1;103(4):461-72. doi: 10.1093/cvr/cvu157. Epub 2014 Jun 19. PMID 24947415
- [Background] Islam MN, Das SR, Emin MT, Wei M, Sun L, Westphalen K, Rowlands DJ, Quadri SK, Bhattacharya S, Bhattacharya J. Mitochondrial transfer from bone-marrow-derived stromal cells to pulmonary alveoli protects against acute lung injury. Nat Med. 2012 Apr 15;18(5):759-65. doi: 10.1038/nm.2736. PMID 22504485
- [Background] Eirin A, Zhu XY, Ebrahimi B, Krier JD, Riester SM, van Wijnen AJ, Lerman A, Lerman LO. Intrarenal Delivery of Mesenchymal Stem Cells and Endothelial Progenitor Cells Attenuates Hypertensive Cardiomyopathy in Experimental Renovascular Hypertension. Cell Transplant. 2015;24(10):2041-53. doi: 10.3727/096368914X685582. Epub 2014 Nov 21. PMID 25420012
- [Background] Katsuno T, Ozaki T, Saka Y, Furuhashi K, Kim H, Yasuda K, Yamamoto T, Sato W, Tsuboi N, Mizuno M, Ito Y, Imai E, Matsuo S, Maruyama S. Low serum cultured adipose tissue-derived stromal cells ameliorate acute kidney injury in rats. Cell Transplant. 2013;22(2):287-97. doi: 10.3727/096368912X655019. Epub 2012 Sep 7. PMID 22963874
- [Background] Donizetti-Oliveira C, Semedo P, Burgos-Silva M, Cenedeze MA, Malheiros DM, Reis MA, Pacheco-Silva A, Camara NO. Adipose tissue-derived stem cell treatment prevents renal disease progression. Cell Transplant. 2012;21(8):1727-41. doi: 10.3727/096368911X623925. Epub 2012 Feb 2. PMID 22305061
- [Background] Zhu XY, Ebrahimi B, Eirin A, Woollard JR, Tang H, Jordan KL, Ofori M, Saad A, Herrmann SM, Dietz AB, Textor SC, Lerman A, Lerman LO. Renal Vein Levels of MicroRNA-26a Are Lower in the Poststenotic Kidney. J Am Soc Nephrol. 2015 Jun;26(6):1378-88. doi: 10.1681/ASN.2014030248. Epub 2014 Sep 30. PMID 25270070
- [Background] Takasato M, Er PX, Chiu HS, Maier B, Baillie GJ, Ferguson C, Parton RG, Wolvetang EJ, Roost MS, Chuva de Sousa Lopes SM, Little MH. Kidney organoids from human iPS cells contain multiple lineages and model human nephrogenesis. Nature. 2015 Oct 22;526(7574):564-8. doi: 10.1038/nature15695. Epub 2015 Oct 7. PMID 26444236
- [Background] Liu Y. Cellular and molecular mechanisms of renal fibrosis. Nat Rev Nephrol. 2011 Oct 18;7(12):684-96. doi: 10.1038/nrneph.2011.149. PMID 22009250
- [Background] Sun D, Eirin A, Ebrahimi B, Textor SC, Lerman A, Lerman LO. Early atherosclerosis aggravates renal microvascular loss and fibrosis in swine renal artery stenosis. J Am Soc Hypertens. 2016 Apr;10(4):325-35. doi: 10.1016/j.jash.2016.01.019. Epub 2016 Jan 28. PMID 26879682
- [Background] Ma YY, Sun D, Li J, Yin ZC. Transplantation of endothelial progenitor cells alleviates renal interstitial fibrosis in a mouse model of unilateral ureteral obstruction. Life Sci. 2010 May 22;86(21-22):798-807. doi: 10.1016/j.lfs.2010.03.013. Epub 2010 Mar 20. PMID 20331991
- [Background] Sun D, Bu L, Liu C, Yin Z, Zhou X, Li X, Xiao A. Therapeutic effects of human amniotic fluid-derived stem cells on renal interstitial fibrosis in a murine model of unilateral ureteral obstruction. PLoS One. 2013 May 28;8(5):e65042. doi: 10.1371/journal.pone.0065042. Print 2013. PMID 23724119
- [Background] Eirin A, Zhu XY, Krier JD, Tang H, Jordan KL, Grande JP, Lerman A, Textor SC, Lerman LO. Adipose tissue-derived mesenchymal stem cells improve revascularization outcomes to restore renal function in swine atherosclerotic renal artery stenosis. Stem Cells. 2012 May;30(5):1030-41. doi: 10.1002/stem.1047. PMID 22290832
- [Background] Zhu XY, Urbieta-Caceres V, Krier JD, Textor SC, Lerman A, Lerman LO. Mesenchymal stem cells and endothelial progenitor cells decrease renal injury in experimental swine renal artery stenosis through different mechanisms. Stem Cells. 2013 Jan;31(1):117-25. doi: 10.1002/stem.1263. PMID 23097349
- [Background] Roemeling-van Rhijn M, Reinders ME, de Klein A, Douben H, Korevaar SS, Mensah FK, Dor FJ, IJzermans JN, Betjes MG, Baan CC, Weimar W, Hoogduijn MJ. Mesenchymal stem cells derived from adipose tissue are not affected by renal disease. Kidney Int. 2012 Oct;82(7):748-58. doi: 10.1038/ki.2012.187. Epub 2012 Jun 13. PMID 22695328
- [Background] Warner L, Glockner JF, Woollard J, Textor SC, Romero JC, Lerman LO. Determinations of renal cortical and medullary oxygenation using blood oxygen level-dependent magnetic resonance imaging and selective diuretics. Invest Radiol. 2011 Jan;46(1):41-7. doi: 10.1097/RLI.0b013e3181f0213f. PMID 20856128
- [Background] Ebrahimi B, Gloviczki M, Woollard JR, Crane JA, Textor SC, Lerman LO. Compartmental analysis of renal BOLD MRI data: introduction and validation. Invest Radiol. 2012 Mar;47(3):175-82. doi: 10.1097/RLI.0b013e318234e75b. PMID 22183077
- [Background] Saad A, Crane J, Glockner JF, Herrmann SM, Friedman H, Ebrahimi B, Lerman LO, Textor SC. Human renovascular disease: estimating fractional tissue hypoxia to analyze blood oxygen level-dependent MR. Radiology. 2013 Sep;268(3):770-8. doi: 10.1148/radiol.13122234. Epub 2013 Jun 20. PMID 23788716
- [Background] Li Q, Li J, Zhang L, Chen Y, Zhang M, Yan F. Diffusion-weighted imaging in assessing renal pathology of chronic kidney disease: A preliminary clinical study. Eur J Radiol. 2014 May;83(5):756-62. doi: 10.1016/j.ejrad.2014.01.024. Epub 2014 Feb 7. PMID 24581595
- [Background] Inoue T, Kozawa E, Okada H, Inukai K, Watanabe S, Kikuta T, Watanabe Y, Takenaka T, Katayama S, Tanaka J, Suzuki H. Noninvasive evaluation of kidney hypoxia and fibrosis using magnetic resonance imaging. J Am Soc Nephrol. 2011 Aug;22(8):1429-34. doi: 10.1681/ASN.2010111143. Epub 2011 Jul 14. PMID 21757771